CLINICAL TRIAL: NCT02590328
Title: Generalized Neonatal Screening for Severe Combined Immunodeficiencies (SCID) by Quantification of TRECs
Brief Title: Neonatal Screening of Severe Combined Immunodeficiencies
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jinqiao Sun, Professor, Children's Hospital of Fudan University
Other Study IDs: NSSCID
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-01

CONDITIONS: Severe Combined Immunodeficiency; Neonatal Screening
Keywords: Neonatal Screening; Severe Combined Immunodeficiency; Immunologic Deficiency Syndromes; DNA Repair-Deficiency Disorders; T-cell Receptor Excision Circle
MeSH Terms: conditions — Severe Combined Immunodeficiency; Immunologic Deficiency Syndromes; DNA Repair-Deficiency Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Some drops of blood stored on the neonatal screening card (Guthrie card) as a source of DNA to screening. Samples is performed after parents' information and consent. The card drawn for the protocol will follow the usual network except that the test for quantifying TRECs will be realized to determine the presence of SCID.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Screened patients: SCID screening: some drops of blood are placed on a second Guthrie card when current screening is performed after parents' information and consent. The card drawn for the protocol will follow the usual network except that the test for quantifying TRECs will be realized to determine the presence of SCID.

SUMMARY:
The goal of the proposed research is to observe the prevalence and establish the validity of a newborn screening method for severe combined immunodeficiency (SCID). The assay to be used is developed on the basis of PCR quantification of T-cell receptor excision circles (TRECs) that is absent in SCID patients, thus correlating with the disease.

DETAILED DESCRIPTION:
Severe combined Immunodeficiencies (SCID) are a group of inherited diseases of the immune system by characterized profound abnormalities of B and T cell development. Infants with SCID require prompt clinical response to prevent life threatening infection and studies show significantly improved survival in babies Diagnosed at birth as a result of previous family history. SCID follows criteria for population based newborn screening since it is asymptomatic at birth and fatal within the first year of life, the confirmation of the disease is easy, there is a curative treatment, and it is known that early stem cell transplantation improves survival.To show that early diagnosis of SCID with a TREC screening assay can warrant timely treatment of the disease and avoid life-threatening infections on patients. Babies with SCID are unable to fight infections. They become severely ill in their first months of life and do not survive unless their immune systems can be restored. SCID can be treated by bone marrow transplant if recognized early. We undertake the task of newborn screening in the whole region of Shanghai, So the newborn screening test to be employed in this study is designed to diagnose SCID before infections occur. Through this study, we hope to confirm the prevalence of SCID in China and the benefits of newborn screening for early diagnosis of SCID.

Quantification of TRECs (T-cell receptor excision circles) in DNA extracted from Guthrie samples is a sensitive screening test for Specific and SCID. TRECs are small-circle DNA molecules which are by-products of T cell maturation in the thymus, and their numbers reflect the number of recently emigrated T-cells from the thymus. Since all infants with SCID have a profound decrease in T-lymphocytes no matter what gene mutations are involved, logically the number of TRECs present in blood collected via dried blood spots 1-2 days post delivery on SCID babies should be very low when compared with healthy newborns. The TREC assay includes DNA extraction from a 3 mm punch of dried blood specimen in a 96-well plate format. The extracted DNA undergoes Real-time qPCR procedure on 7900 HT Fast Real-time PCR System (ABI). The TREC copy number is calculated relative to a standard curve generated from serially diluted plasmids which contain a known number of TREC. The investigators propose in this study to perform a neonatal screening of SCID, in a population of 200,000 babies over a period of three years. The investigators propose to study the incidence of SCID, mortality & rate of disability, clinical utility and SCID screening to demonstrate that could result in a broad benefit to individuals detected, making screening relatively efforts in spite of the low incidence of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. No more than 28 days old
2. Newborns who was born in Shanghai and in 2016 to 2020
3. Blood sample card was collected in 72 hours after birth

Exclusion Criteria:

1. Lack of parental consent
2. Sample card was damaged

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Screening newborns will be selected from all cooperative hospitals of Neonatal Screening Programme in Shanghai who was born from 2016 to 2020.
Sampling Method: Non-Probability Sample
Enrollment: 180000 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
prevalence of SCID | At 28 days after birth

SECONDARY OUTCOMES:
Number of detected SCID patients | At 28 days after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kobrynski L. Newborn screening for severe combined immune deficiency (technical and political aspects). Curr Opin Allergy Clin Immunol. 2015 Dec;15(6):539-46. doi: 10.1097/ACI.0000000000000221. PMID 26485096
- [Background] de Pagter AP, Bredius RG, Kuijpers TW, Tramper J, van der Burg M, van Montfrans J, Driessen GJ; Dutch Working Party for Immunodeficiencies. Overview of 15-year severe combined immunodeficiency in the Netherlands: towards newborn blood spot screening. Eur J Pediatr. 2015 Sep;174(9):1183-8. doi: 10.1007/s00431-015-2518-4. Epub 2015 Apr 1. PMID 25875249
- [Background] Rozmus J, Junker A, Thibodeau ML, Grenier D, Turvey SE, Yacoub W, Embree J, Haddad E, Langley JM, Ramsingh RM, Singh VA, Long R, Schultz KR. Severe combined immunodeficiency (SCID) in Canadian children: a national surveillance study. J Clin Immunol. 2013 Nov;33(8):1310-6. doi: 10.1007/s10875-013-9952-8. PMID 24122030
- [Background] Puck JM, Routes J, Filipovich AH, Sullivan K. Expert commentary: practical issues in newborn screening for severe combined immune deficiency (SCID). J Clin Immunol. 2012 Feb;32(1):36-8. doi: 10.1007/s10875-011-9598-3. Epub 2011 Oct 20. No abstract available. PMID 22012274
- [Background] Burroughs L, Woolfrey A. Hematopoietic cell transplantation for treatment of primary immune deficiencies. Cell Ther Transplant. 2010 Aug 31;2(8):10.3205/ctt-2010-en-000077.01. doi: 10.3205/ctt-2010-en-000077.01. PMID 21152385
- [Background] Puck JM. Neonatal screening for severe combined immune deficiency. Curr Opin Allergy Clin Immunol. 2007 Dec;7(6):522-7. doi: 10.1097/ACI.0b013e3282f14a2a. PMID 17989529
- [Background] Puck JM; SCID Newborn Screening Working Group. Population-based newborn screening for severe combined immunodeficiency: steps toward implementation. J Allergy Clin Immunol. 2007 Oct;120(4):760-8. doi: 10.1016/j.jaci.2007.08.043. PMID 17931561
- [Background] de Silva R, Gunasena S, Ratnayake D, Wickremesinghe GD, Kumarasiri CD, Pushpakumara BA, Deshpande J, Kahn AL, Sutter RW. Prevalence of prolonged and chronic poliovirus excretion among persons with primary immune deficiency disorders in Sri Lanka. Vaccine. 2012 Dec 14;30(52):7561-5. doi: 10.1016/j.vaccine.2012.10.035. Epub 2012 Oct 22. PMID 23099333